CLINICAL TRIAL: NCT02669576
Title: Mind-Body Medicine Day Care Clinic in Breast Cancer Patients Undergoing Endocrine Therapy: A Randomized Controlled Trial.
Brief Title: Mind-Body Medicine Day Care Clinic in Breast Cancer Patients Undergoing Endocrine Therapy
Acronym: ENDOTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Postdoctoral Research Fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-6578-BO
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; meopausal syptoms; mind body medecine; yoga; acupuncture
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind body medicine day care clinic (Experimental): Patients recieve an 11-week mind body day care clinic including elements of mindfullness based stress reduction (MBSR), yoga, acupuncture, education
  Interventions: Behavioral: Mind body medicine day care clinic
- Usual care (Other): Patients continue usual care by their practitioner
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Mind body medicine day care clinic — Patients recieve an 11-week mind body day care clinic including elements of mindfullness based stress reduction (MBSR), yoga, acupuncture, education
  Arms: Mind body medicine day care clinic
Other: Usual care — Patients continue usual care by their practitioner
  Arms: Usual care

SUMMARY:
This randomized controlled trial aims to investigate the effectiveness of a mind body day care clinic program of breast cancer patients undergoing endocrine therapy.

DETAILED DESCRIPTION:
Breast cancer patients undergoing endocrine therapy are often suffering from side effects. This randomized controlled trial analyzes the effects of an 11-week day care clinic group program including mind body medical elements (yoga, relaxation, meditation, education) and acupuncture in breast cancer patients with menopausal symptoms under endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosed breast cancer (Stage I-III), no metastases
* Current endocrine therapy (minimum 3 months)
* Score of 9 or greater on the Menopausal Rating Scale (MRS)
* Signed informed consent

Exclusion Criteria:

* Severe other somatic or psychiatric comorbidity
* Pregnancy
* Planned or existing chemotherapy, radiation or other cure treatment
* Participation in other clinical studies with behaviour-oriented, psychological or compementary medicine intervention.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Menopausal symptoms | week 11
  Menopause Rating Scale (MRS)

SECONDARY OUTCOMES:
General health-related quality of life | week 11
  Functional Assessment of Cancer Therapy - General Questionaire (FACT-G)
Spiritual health-related quality of life | week 11
  Functional Assessment of Cancer Therapy - Spirutual Subscale (FACT-SP)
Fatigue | week 11
  Functional Assessment of Cancer Therapy - Fatigue Subscale (FACT-F)
Mental wellbeing | week 11
  Hospital Anxiety and Depression Scale (HADS)
Stress | week 11
  Perceived Stress Scale (PSS)
Compliance | week 11
  Medication Adherence Report Scale (MARS)
Adverse events | week 11
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Menopausal smptoms | week 23
  Menopause Rating Scale (MRS)
Genaeral health-related quality of life | week 23
  Functional Assessment of Cancer Therapy - General Questionaire (FACT-G)
Spiritual health-related quality of life | week 23
  Functional Assessment of Cancer Therapy - Spirutual Subscale (FACT-SP)
Fatigue | week 23
  Functional Assessment of Cancer Therapy - Fatigue Subscale (FACT-F)
Mental wellbeing | week 23
  Hospital Anxiety and Depression Scale (HADS)
Stress | week 23
  Perceived Stress Scale (PSS)
Compliance | week 23
  Medication Adherence Report Scale (MARS)
Adverse Events | week 23
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
Mindfulness | week 11
  Conscious Presence and Self Control Scale (CPSC)
Social Support | week 11
  Berlin Social Support Scale (BSSS)
Expectation | week 0
  Visual Analogue Scale (VAS)
Statisfaction | week 11
  Client Satisfaction Questionnaire (CSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — Center for Integrative Medicine and Health, University Hospital Essen, University of Duisburg-Essen
Locations (1):
- Evang. Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No